CLINICAL TRIAL: NCT07012291
Title: Multi-site Clinical Performance Evaluation of Native Whole Blood Samples of Patients on Direct Oral Anticoagulants (DOACs) With the Perosphere ClotChek™ Coagulometer
Brief Title: Clinical Performance Evaluation of Native Whole Blood Samples of Patients on DOACs With the Perosphere ClotChek™
Status: Recruiting | Type: Observational
Sponsor: Perosphere Technologies Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-01-03-001
Record Dates: First submitted 2025-05-19; First posted 2025-06-10 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-06

CONDITIONS: Coagulation
MeSH Terms: conditions — Thrombosis | interventions — Whole Blood Coagulation Time

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Whole Blood Clotting Time — Fresh whole blood samples from patients on rivaroxaban or apixaban taken at various times during the day to obtain samples from DOAC patients that represent the entire analytical range to the extent possible, as opposed to a strict "trough/peak" testing schedule.
Device: Whole Blood Clotting Time — Fresh whole blood samples, non-citrated, are drawn and loaded onto a cuvette free of any biological reagents, to obtain a whole blood clotting time value.

SUMMARY:
The Perosphere ClotChek™ system consists of a hand-held, battery-operated blood coagulation instrument and disposable test cuvettes for use at the point-of-care (POC). The instrument performs a whole blood clotting time (WBCT) test using freshly drawn, non-citrated whole blood. The purpose of the present study is to characterize the performance of the Perosphere ClotChek™ as a quantitative measurement of the WBCT in patients taking one of the following Direct Oral Anticoagulants (DOACs), rivaroxaban or apixaban.

ELIGIBILITY:
Inclusion Criteria:

* Be informed of the nature of the study and provide written informed consent before any study-specific procedures are performed.
* Be 18- to 80-years-of-age, inclusive, at time of consent.
* Have suitable venous access for at least a single venipuncture.
* Eligible patients on anticoagulants must have taken their prescribed anticoagulant regularly at least for one month prior to study participation for inclusion
* Eligible patients on anticoagulants must have been on their anticoagulant therapy for at least one month.

Exclusion Criteria:

* Have a personal or family history of clotting disorder or hematologic abnormality, such as excessive bleeding, joint hematoma, thrombovascular disease, thrombocytopenia, or any chronic condition requiring treatment with transfusions, other than the condition for which a DOAC was prescribed.
* Have a history of unexplained syncope.
* Have a history within six months prior to Screening of peptic ulcer or gastrointestinal bleeding (including hematemesis, melena, or rectal bleeding).
* Consume more than five cigarettes per day.
* If female, have a history of excessive or dysfunctional uterine bleeding (unless the subject had a subsequent hysterectomy).
* If female, be pregnant, breastfeeding, or planning to become pregnant during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on rivaroxaban or apixaban between the ages of 18 and 80 years old.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Differentiating DOAC patients taking rivaroxaban or apixaban from normal control patients, via measurement of their whole blood clotting time. | Day 1

SECONDARY OUTCOMES:
To characterize performance of the ClotChek™ device via whole blood clotting time measurement within clinically relevant patient subgroups (eg renal or hepatic impairment). | Day 1

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Perosphere Technologies Inc, Danbury, Connecticut
  - Perosphere Technologies Inc, Rockville, Maryland
  - Eastern Vascular Associates, Denville, New Jersey
  - Bassett Research Institute - Center for Clinical Research, Cooperstown, New York

IPD SHARING:
Plan to Share IPD: No